CLINICAL TRIAL: NCT05799027
Title: Raman Spectroscopic Analysis of Bronchoscopic Biopsy for Diagnosing Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Principal Investigator, China-Japan Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-NHLHCRF-LX-01-0201-05
Record Dates: First submitted 2023-03-08; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Raman spectrum analysis (Experimental): The bronchoscopic biopsy sample of patients with visible lesions in the airway would undergo raman spectrum analysis.
  Interventions: Diagnostic Test: Raman spectrum

INTERVENTIONS:
Diagnostic Test: Raman spectrum — The bronchoscopic biopsy sample of patients with visible lesions in the airway would undergo raman spectrum analysis.

SUMMARY:
The goal of this clinical trial is to evaluate raman spectroscopic analysis of bronchoscopic biopsy for diagnosing lung cancer in visible lesions in the airway. The main question it aims to answer are: the diagnostic efficacy raman spectroscopic analysis of bronchoscopic biopsy for diagnosing lung cancer.

The bronchoscopic biopsy sample of patients with visible lesions in the airway would undergo raman spectrum analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who plan to undergo bronchoscopic biopsy or EBUS-TBNA
* Visible intratracheal lesions under bronchoscope
* Non-visible lesions suspected of lung cancer

Exclusion Criteria:

* The patient could not tolerate further examination aimed at clarifying the cause of the disease or refused to accept further examination aimed at clarifying the cause of the disease due to poor general condition, serious organ dysfunction, etc
* The patient has no definite diagnosis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-03-31 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
To establish the sensitivities and specificities of Raman spectroscopic analysis of bronchoscopic biopsy for lung cancer. | 7 days after the biopsy
  The diagnosis would be confirmed according to the pathological results.